CLINICAL TRIAL: NCT06167408
Title: Identifying Factors Influencing In-Hospital Relapse in Pemphigus Patients: A Retrospective Study
Brief Title: Identifying Factors Influencing In-Hospital Relapse in Pemphigus Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hanyi Wu, doctor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 20231130
Record Dates: First submitted 2023-11-30; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Pemphigus Vulgaris
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pemphigus patients in the First Affiliated Hospital of Chongqing Medical University

SUMMARY:
The objective of this retrospective study was to investigate the factors influencing in-hospital relapse during acute episodes of pemphigus, an autoimmune blistering disease characterized by self-antibodies targeting desmogleins. The study included 96 pemphigus patients hospitalized in China between January 2014 and December 2020. The primary questions addressed by the study were:

What are the risk factors associated with in-hospital relapse during acute episodes of pemphigus? Participants in the study underwent a retrospective analysis using univariate and multivariate Cox regression analysis to identify and understand the various risk factors contributing to in-hospital relapse. This research aimed to contribute valuable insights into the factors influencing the course of pemphigus, providing crucial information for better management and treatment strategies.

DETAILED DESCRIPTION:
This retrospective study conducted in China between January 2014 and December 2020 aimed to comprehensively examine factors influencing in-hospital relapse during acute episodes of pemphigus, an autoimmune blistering disease characterized by self-antibodies targeting desmogleins-essential cell adhesion molecules. The study enrolled 96 pemphigus patients who were hospitalized during acute episodes.

Research Questions:

Primary Question:

What are the identifiable risk factors associated with in-hospital relapse in pemphigus patients during acute episodes?

Methods:

Study Type: Retrospective Observational Study Participant Population: 96 pemphigus patients hospitalized in China Duration: January 2014 to December 2020

Main Tasks:

Data Collection:

Retrospective analysis of medical records and clinical data of pemphigus patients during acute hospitalizations.

Identification of demographic information, clinical characteristics, and treatment modalities.

Risk Factor Determination:

Univariate and multivariate Cox regression analysis employed to assess potential risk factors.

Variables considered included demographic factors, disease severity, and specific treatment regimens.

Outcome Measurement:

Identification of in-hospital relapse as the primary outcome. Correlation of relapse occurrence with the identified risk factors.

Results:

Key Findings:

Identification of specific risk factors contributing to in-hospital relapse in pemphigus patients.

Quantification of the impact of demographic and clinical variables on relapse probability.

Significance:

Clinical Implications:

Contribution of valuable insights for clinicians in predicting and managing in-hospital relapse in pemphigus patients.

Informing treatment strategies based on identified risk factors.

Research Contribution:

Expansion of understanding regarding the course and management of pemphigus. Providing a foundation for future prospective studies and the development of targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* inpatients.
* Pathologic diagnosis of pemphigus.

Exclusion Criteria:

* Patients hospitalized for cyclophosphamide shock therapy only.
* Patients who did not recover and were discharged due to personal reasons.

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included 96 patients diagnosed with pemphigus who received inpatient treatment at the First Affiliated Hospital of Chongqing Medical University between January 1st, 2014, and December 31st, 2020. The inclusion criteria covered both initial and follow-up cases, without age or sex restrictions. Diagnosis was confirmed through pathological biopsy, classifying pemphigus into different types. Patients underwent routine assessments, received various treatments, and were monitored for complications during hospitalization. Ten patients with multiple hospitalizations for cyclophosphamide pulse therapy and three patients not recovering were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
in-hospitalization relapse | through hospitalization (Up to 1 month)
  the occurrence of in-hospital relapse among pemphigus patients during acute episodes

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated hospital of Chongqing Medical University, Chongqing, Yuzhong District, China

IPD SHARING:
Plan to Share IPD: No